CLINICAL TRIAL: NCT04679740
Title: RMS (Resorbable Magnesium Scaffolds) Registry
Brief Title: Resorbable Magnesium Scaffolds Registry
Status: Recruiting | Type: Observational
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C1908
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease
Keywords: Registry; Magmaris; Coronary Artery Disease; PCI; Resorbable Magnesium Scaffolds; Freesolve
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Magmaris — MAGMARIS is indicated for improving luminal diameter in the treatment of de novo native coronary artery lesions in patients with symptomatic coronary artery disease. The reference vessel diameter should closely match the scaffold nominal diameter. The treated lesion length should be less than the nominal scaffold length.
  Other Names: Magmaris Sirolimus-Eluting Resorbable Coronary Magnesium Scaffold
Device: Freesolve — Freesolve is indicated for improving luminal diameter in the treatment of de novo native coronary artery lesions in patients with symptomatic coronary artery disease. The reference vessel diameter should closely match the scaffold nominal diameter. The treated lesion length should be less than the nominal scaffold length.
  Other Names: Freesolve Sirolimus-Eluting Coronary Resorbable Magnesium Scaffold (RMS) System

SUMMARY:
The registry follows the ESC/EACTS guideline and further investigates the clinical performance and short-term safety of RMS (Resorbable Magnesium Scaffolds) in a real world setting within the scope of its intended use without further (medical related) exclusion criteria according to their respective instructions for use (IFU).

ELIGIBILITY:
Inclusion Criteria:

* According to the IFU

Exclusion Criteria:

* According to the IFU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic coronary artery disease needing the treatment of de novo native coronary artery lesions
Sampling Method: Non-Probability Sample
Enrollment: 1106 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  The primary endpoint will be Target Lesion Failure (TLF) at 12 months. TLF is a composite of Cardiac Death, Target Vessel Q-wave or non-Q wave MI, or clinically driven Target Lesion Revascularization (TLR).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Galli, MD, Principal Investigator — Centro Cardiologico Monzino
Locations (13):
- Cairns Hospital, Cairns, Australia
- Germany (5):
  - Heart Center Segeberger Kliniken, Bad Segeberg
  - Krankenhaus Buchholz, Buchholz
  - Klinikum Westfalen, Knappschaft KH, Dortmund
  - Klinikum Herford, Herford
  - Herz-und Gefäßzentrum Oberallgäu-Kempten, Kempten
- Centro Cardiologico Monzino, Milan, Lombardy, Italy
- Daugavpils Regional Hospital, Daugavpils, Latvia
- 1 Wojskowy Szpital Kliniczny z Poliklinika SPZOZ w Lublinie, Lublin, Poland
- SUSCCH Banska Bystrica, Banská Bystrica, Slovakia
- Switzerland (3):
  - Lindenhofspital, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Solothurner Spitäler AG, Olten

IPD SHARING:
Plan to Share IPD: No
The primary outcome data will be shared after the publication of it.